CLINICAL TRIAL: NCT01235858
Title: Responding to the ASRA (American Society of Regional Anesthesia) Challenge - Should Gowning be the Standard of Practice for Epidural Anesthesia: A Randomized Control Trial
Brief Title: Aseptic Techniques During Epidural Analgesia in the Labor Floor
Acronym: EAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Principal Investigator, Dr. Naveed Siddiqui, Principal Investigator, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EAS-2009
Record Dates: First submitted 2010-09-27; First posted 2010-11-08 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2011-07

CONDITIONS: Pregnancy
Keywords: Epidural analgesia; Epidural anesthesia labor; Aseptic technique; gown; no gown

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gown group (Other): Anesthesiologists wearing sterile gown for epidural insertion
  Interventions: Procedure: wearing of sterile gowns
- No Gown group (Other): Anesthesiologists not wearing gown for epidural insertion
  Interventions: Procedure: No gown

INTERVENTIONS:
Procedure: wearing of sterile gowns — Anesthesiologists wearing sterile gown for epidural insertion
  Other Names: Sterile gowns
  Arms: Gown group
Procedure: No gown — Anesthesiologists not wearing sterile gown for epidural insertion
  Arms: No Gown group

SUMMARY:
There is an increasing trend in the incidence of infection related to epidural anesthesia. This could be related to methods of aseptic technique as adopted by the anesthesiologist during the performance of the procedure.

The purpose of this study is to compare two methods of aseptic technique for labor epidural insertion; a "conventional" method without wearing a sterile gown (free from living germs or microorganisms) versus strict aseptic method with wearing of sterile gowns.

It is our belief that there will be an increased contamination of epidural equipment and colonization of epidural catheter, secondary to bacterial fallout from the operators' bare hands in the group not wearing the sterile gowns.

DETAILED DESCRIPTION:
At the present time there is no accepted standard for aseptic technique during insertion of an epidural catheter on the labor floor and what is considered to be essential is controversial. Recognizing this, the American Society of Regional Anesthesia (ASRA), the leading authority on regional anesthesia, established a task force to examine and establish guidelines for aseptic practice. Their findings highlighted the lack of good quality studies to support specific recommendations. This is especially true in regards to the use of sterile gowns during the performance of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women requesting epidural analgesia

Exclusion Criteria:

* Patients who have fever requiring antibiotics
* Patients who have received antibiotics in or within the previous 48 hours of labor
* Immuno-compromised patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Growth of microbial organisms on operators forearm, agar plate (working area) and proximal and distal tip of the epidural catheter. | one and one half year

SECONDARY OUTCOMES:
length of epidural catheterization and positive culture | one year and a half

CONTACTS AND LOCATIONS:
Overall Officials: Naveed T Siddiqui, MD, Principal Investigator — Department of Anesthesia and Pain Management Mount Sinai Hospital, Toronto,Canada
Locations (1):
- Department of Anesthesia Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Siddiqui NT, Davies S, McGeer A, Carvalho JC, Friedman Z. The effect of gowning on labor epidural catheter colonization rate: a randomized controlled trial. Reg Anesth Pain Med. 2014 Nov-Dec;39(6):520-4. doi: 10.1097/AAP.0000000000000171. PMID 25304478